CLINICAL TRIAL: NCT06673082
Title: Impact of Zinc as a New Adjuvant Therapy for Cow Milk Protein Allergy in Children, A Randomized Controlled Trial
Brief Title: Impact of Zinc as a New Adjuvant Therapy for Cow Milk Protein Allergy in Children.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Arwa Ahmed, pediatric specialist, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: zinc in cow milk allergy; Arwa (Other: self funding)
Record Dates: First submitted 2024-10-22; First posted 2024-11-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: Cow Milk Protein Allergy
Keywords: Zinc; Cow Milk Protein Allergy; COMISS; SCORAD

STUDY DESIGN:
Intervention Model Description: one group will receive oral Zinc therapy while the other group will recieve placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional group (Experimental): Oral Zinc will be supplemented to the interventional group on a dose of 30 mg elemental zinc/day.
  Interventions: Drug: Oral zinc supplementation
- control group (Placebo Comparator): oral placebo identical to Zinc inappearance and packaging
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral zinc supplementation — Oral Zinc will be supplemented to the interventional group on a dose of 30 mg elemental zinc/day.
  Arms: interventional group
Other: Placebo — Oral
  Arms: control group

SUMMARY:
Children presented with manifestations of Cow Milk Protein Allergy will be enrolled for Cow Milk -related Symptoms Score (CoMiSS assessment). Detailed History, nutritional and clinical examination will be done to fulfill items of CoMiSS. Children will be randomly allocated to two groups. Oral Zinc will be supplemented to the interventional group. CoMiSS will be recorded at the baseline and weekly till 4 weeks. Then Oral Food Challenge (OFC) will be done to confirm the diagnosis and CoMiSS assessment will be recorded again to see if Zinc has any modulatory effect on reappearance of symptoms. The people administering the intervention, the people assessing the outcomes, the patients and their caregivers will all be blinded to the type of treatment.

Children who will be presented with skin manifestation will be assessed by Severity Scoring of Atopic Dermatitis Index (SCORAD score) once diagnosed and weekly till 4 weeks after zinc supplementation to see if Zinc has any modulatory effect.

DETAILED DESCRIPTION:
Children who will be presented with manifestations of Cow Milk Protein Allergy will be enrolled in the study for Cow Milk -related Symptoms Score (CoMiSS) assessment.

Detailed History, nutritional and clinical examination will be done to fulfill items of CoMiSS including skin manifestations as eczema , respiratory manifestations, GIT manifestations as constipation or diarrhea including Bristol scale and regurgitations and duration of crying .

Children will be randomly allocated to two groups. Randomization will be done using GraphPad QuickCalcs software to allocate into either the interventional or control group. Oral Zinc will be supplemented to the interventional group on adose of 30 mg elemental zinc/day.

CoMiSS will be recorded at the baseline and weekly till 4 weeks. Then Oral Food Challenge (OFC) will be done to confirm the diagnosis and CoMiSS assessment will be recorded againto see if Zinc has any modulatory effect on reappearance of symptoms. The people administering the intervention, the people assessing the outcomes, the patients and their caregivers will all be blinded to the type of treatment.

Children who will be presented with skin manifestation will be assessed by Severity Scoring of Atopic Dermatitis Index (SCORAD score) once diagnosed and weekly till 4 weeks after zinc supplementation to see if Zinc has any modulatory effect.

ELIGIBILITY:
Inclusion Criteria:

Children suspected to have Cow Milk Protein Allergy using Cow's Milk-relatedSymptoms Score with a Score more than12 Age less than 12 years old both sexes Whose parents approved to be enrolled in the study

Exclusion Criteria:

Children with Comorbidities that may affect the duration of treatment as dysphagia.

History of Severe allergic reaction that required hospital admission as Ora Food Challenge is expectedto be delayed in these patients.

-Multiple Food Allergies

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
COMISS(Cow Milk Related symptom Score) | 2 weeks
  Evaluate the degree of change in COMISS Sc0re(Cow Milk Related symptom Score) between the interventional group and control group The COMISS Score ranges from 0 to 33. Each symptom has a maximal score of six,exception of respiratory symptoms(maximal score of three).
  a cut-off value>12 was selected as the criterion to pick up infant at risk of Cow Milk Allergy . A score of 12 requires the presence of at least two severe symptoms and a score higher than10 requires the precense of at least three symptoms and the involvement of two organ systems

SECONDARY OUTCOMES:
COMISS (Cow Milk Related Symptom Score)and SCORAD (Severity Scoring of Atopic Dermatitis index) | 4 Weeks
  1. Degree of change clinicaiiy by SCORAD (Severity Scoring of Atopic Dermatitis index) between the intervention and control group upon Zinc adminstration.
     SCORAD is a clinical tool used to assess the extent and severity of eczema, To determine extent by is the 'rule of nine': 9% for the head and neck, each arm, the front and back of each leg, the four trunk quadrants, and 1% for the genitalia, The intensity part of the index consists of six items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness. Each item can be graded on a scale 0-3 pruritus and sleeplessness (0-10)for each, SCORAD score range is between 0 and 103 points and defines three classes of AD severity (. mild if SCORAD <25, moderate if 25 ≤ SCORAD ≤ 50 and severe if SCORAD > 50.
  2. The Change in the degree of improvement between the interventional and control group based on COMISS score at 1,2, 3, and 4 weeks.
  2.Time to improvement of COMISS score below 12 in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Abdelaziz, Professor of Pediatrics, Principal Investigator — Cairo University; Dalia Sayed Mosallam, Professor of Pediatrics, Principal Investigator — Cairo University; Hoda Atef Abdel Sattar, Lecturer of Pediatrics, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine-Cairo universty, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No